CLINICAL TRIAL: NCT00420108
Title: Comparing ICD Device Diagnostics to Hospitalized Heart Failure Patient Symptoms and Physician Opinion on Discharge Readiness
Brief Title: Optivol Diagnostic Data for Discharge in Heart Failure
Acronym: 3DHF
Status: Completed | Type: Observational
Sponsor: Thomas Jefferson University (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Office of Research Administration, Thomas Jefferson University
Other Study IDs: 06U.232
Record Dates: First submitted 2007-01-08; First posted 2007-01-09 (Estimated); Last update posted 2010-08-20 (Estimated); Status verified 2010-08

CONDITIONS: Heart Failure, Congestive; Cardiac Pacemaker, Artificial
Keywords: Heart Failure, Congestive; Cardiac Pacemaker, Artificial; Ventricular Pressure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — No biospecimens to be retained
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of this study is to evaluate whether the heart rate variability, daily heart rate, and/or intrathoracic impedance recorded by implantable cardiac devices can be used in conjunction with other traditional clinical practice methods to determine if heart failure patients are ready for hospital discharge.

DETAILED DESCRIPTION:
Implantable cardioverter defibrillator (ICD) devices with or without cardiac resynchronization therapy (CRT-D) have the ability to continuously monitor heart rate variability, daily heart rate, and patient activity. Changes in these measures have been associated with heart failure prognosis. In addition, ICD or CRT-D devices also have the ability to measure daily intrathoracic impedance. Previous data have demonstrated that device-based intrathoracic impedance measurements correlate with pulmonary capillary wedge pressure and fluid retention, both of which are common measures of heart failure status. The objective of this study is to evaluate whether the heart rate variability, daily heart rate, and/or intrathoracic impedance can be used in conjunction with other methods to determine if patients are ready for hospital discharge. This will be the first step in potentially developing an inpatient care strategy which includes implantable device data. It is hypothesized that device diagnostic data will identify an appropriate and safe time to discharge patients admitted for worsening heart failure symptoms before usual clinical indicators. More specifically, we hypothesize that device data will "normalize" at least one day prior to the clinical indicators of readiness for discharge and patients discharged prior to "normalization" of the device data will be at greater risk for rehospitalization

ELIGIBILITY:
Inclusion Criteria:

* Patients implanted with a Medtronic InSync Sentry or subsequent FDA-approved Medtronic device with the OptiVol capability for >30 days.
* Anticipated hospitalization stay >48 hours
* Hospitalized patients experiencing worsening heart failure with symptoms of lung/pulmonary congestion.

Exclusion Criteria:

* Anemia - admission hemoglobin <8.0 g/dL
* Patients residing in convalescence center prior to admission or known to be discharged to a convalescence center or hospice, where discharge could be based on bed availability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is hospitalized patients who have an implanted Medtronic device with Optivol capability.
Sampling Method: Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2006-12; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David J Whellan, MD MHS, Principal Investigator — Thomas Jefferson University
Locations (5):
- United States (5):
  - Heartland Health, Saint Joseph, Missouri
  - Cardiovascular Associates of Delaware Valley, Elmer, New Jersey
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania
  - Main Line Health Lankenau Hospital, Wynnewood, Pennsylvania